CLINICAL TRIAL: NCT03273010
Title: The Efficacy of Cyanoacrylate on Palatal Wound Healing and Postoperative Complaints
Brief Title: The Use of Cyanoacrylate on Palatal Wound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Ceren Gökmenoğlu, Assistant Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ordu Uni
Record Dates: First submitted 2017-08-03; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periacryl group (Experimental): Periacryl, a tissue adhesive, was applied on wound surfaces to achieve haemostasis
  Interventions: Procedure: Free gingival graft; Procedure: Cyanoacrylate application
- Control group (Active Comparator): Free gingival graft was harvested from palatal region and left to heal without applying periacryl.
  Interventions: Procedure: Free gingival graft

INTERVENTIONS:
Procedure: Free gingival graft — Free gingival graft was harvested from palatal donor site
Procedure: Cyanoacrylate application — Periacyrl was applied on palatal wounds
  Arms: Periacryl group

SUMMARY:
The palatal donor site of autogenous free gingival grafts significantly influences the patient's morbidity. The purpose of this study was to evaluate the efficacy of cyanoacrylate on palatal wound healing and postoperative complaints.

DETAILED DESCRIPTION:
A total of 35 patients were included in the study. In the test group (19 patient), cyanoacrylate was placed over the palatal wounds; conversely, the 16 control group patients were allowed to heal in a conventional way without cyanoacrylate.

Primary bleeding time, presence of secondary bleeding, postoperative pain and completion of epithelization were assessed following free gingival graft operation. As a result, compared to the control group it was determined that the cyanoacrylate tissue adhesive could reduce the postoperative morbidity and improve the wound healing.

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases
* no coagulation disorders
* no drug intake in the previous 6 months that might effect the periodontal health status
* no pregnancy or lactation
* no smoking habit
* <1 mm attached gingiva width on one or two lower anterior teeth
* Miller Class I- II- III (Miller 1985) with deep gingival recession (˃ 3mm)

Exclusion Criteria:

* Hematologic disorders
* No cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary bleeding time | baseline
  The moment of active blood flow stasis that a clinical photograph could be taken by examiner without need for suction.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 1-7 days after operation
  The changes in postoperative pain level after the operation
Analgesic consumption | 1-7 days after operation
  The changes in the number of painkiller taken to relieve pain after the operation
Completion of epithelization | Once a week for a month after the operation
  The epithelization assessed by the peroxide test